CLINICAL TRIAL: NCT05073588
Title: Effect of Indo-Mediterranean Diet on Hepatic Steatosis and Fibrosis in Overweight Children and Adolescent With Biopsy Proven NAFLD: A Randomised Control Trial
Brief Title: Effect of Indo-Mediterranean Diet on Hepatic Steatosis and Fibrosis in NAFLD Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-NAFLD-01
Record Dates: First submitted 2021-09-17; First posted 2021-10-11 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2022-09

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: NAFLD; Indo-Mediterranean diet; Calorie restricted diet
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Caloric Restriction

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, Single centre Open label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indo Mediterranean diet (Active Comparator): Indian version of Mediterranean diet will be given to NAFLD children
  Interventions: Other: Indo Mediterranean diet
- Calorie restricted Diet (Active Comparator): Diet restricted in calories will be given to NAFLD children
  Interventions: Other: Calorie restricted diet

INTERVENTIONS:
Other: Indo Mediterranean diet — Mediterranean diet has been shown to be effective in NAFLD adult patients. In India, it is very difficult to follow Mediterranean diet, so one group will be given Indianized version of mediterranean diet.
  Arms: Indo Mediterranean diet
Other: Calorie restricted diet — One group will be given diet restricted in calories, which most of the patients follow to lose weight
  Arms: Calorie restricted Diet

SUMMARY:
NAFLD encompasses the entire spectrum of Fatty liver disease in individuals without significant alcohol consumption, ranging from fatty liver to steatohepatitis to cirrhosis. A high prevalence of NAFLD (62.5%) was observed in overweight/obese Indian adolescent. Lifestyle modification consisting of diet, exercise and weight loss has been advocated to treat patients with NAFLD. European association for study of liver (EASL) guidelines recommends that the macronutrient in the diet should be adjusted according to the Mediterranean diet for weight loss. Mediterranean diet helps to decrease hepatic fat by decreasing lipogenesis, fibrogenesis, inflammation, oxidative stress and by increasing fatty acids beta oxidation.There are numerous studies in adults showing benefit of Mediterranean diet in comparison with other diet in NAFLD, but data on children is very limited. There are no studies in pediatrics showing the benefit of diet intervention in Indian NAFLD children. The aim of this study will be to compare the effect of Indo-Mediterranean diet and calorie restricted on hepatic steatosis and fibrosis in Overweight Indian children and adolescent with Biopsy proven NAFLD.

DETAILED DESCRIPTION:
During the last decade, Nonalcoholic fatty liver disease (NAFLD) has become the most common cause of chronic hepatopathies in children and adolescents. NAFLD is considered as the hepatic manifestation of metabolic syndrome (MetS) and is defined as fat accumulation in the liver of patients who do not consume excessive amounts of alcohol. The mechanism of liver injury in NAFLD is considered to be a "Multiple hit process". The first "hit" leads to an increase in liver fat, while the next multiple factors lead to inflammation. In Developed countries, 4 to 11% of the general pediatric population is affected by NAFLD, reaching a rate of 70% among overweight and obese children. Lifestyle modification consisting of diet, exercise and weight loss has been proven to treat patients with NAFLD. Mediterranean diet (MD) has been largely evaluated for its beneficial effects in terms of prevention of obesity and MetS. Mediterranean diet is a nutritional model which has its origins in stated surrounding the Mediterranean Sea. MD patterns may vary among countries and regions owing to the cultural, ethnic, religious and agricultural differences. MD usually consists of eating primarily unrefined cereals, vegetables and fresh fruit, olive oil, nuts; eating fish, white meat, dairy products in moderation; limiting red meat, processed meats and sweets. MD helps to decrease hepatic fat by decreasing lipogenesis, fibrogenesis, inflammation, oxidative stress and by increasing fatty acids beta oxidation. MD is based on compounds, such as polyphenols, vitamins and other biomolecules that have anti inflammatory and antioxidant effects. It also has carotenoids and lycopenes which act as antioxidants. MD is characterized by high Mono unsaturated fatty acids content with a balanced Poly unsaturated fatty acids omega¬6 to omega¬3 ratio due to the abundance of vegetables, legumes, nuts, olive oil and fish (instead of red meats). There are numerous studies in adults showing benefit of Mediterranean diet in comparison with other diet in NAFLD, but data on children is very limited.

There are only two studies in children on the association between NAFLD and Mediterranean diet. Cakir et al first analysed in obese youth the association between MD adherance {as assessed by the Mediterranean diet quality index (KIDMED)} and NAFLD (as diagnosed by ultrasound and /or elevated ALT levels, as well exclusion of other causes of fatty liver). The authors evaluated overweight/obese children with (n=106) and without (n=21) NAFLD, as well as children (n=54) with normal BMI and without known chronic disease.Subjects with a low MD adherence were more likely to present with a higher BMI, though no correlation was found with other parameters including steatosis severity. Another study by Della Corte et al analysed the adherence to MD {as assessed by the Mediterranean diet quality index(KIDMED) score} in 243 overweight/obese youths with and without NAFLD. Of these, 100 underwent live biopsy. Poor adherance to MD was related to severity of liver damage as well as to higher levels of C-reactive Protein, Insulin and Homeostatic Model Assessment of Insulin Resistance (HOMA IR) values, thus suggesting increased inflammatory potential of unhealthy diets. In the Indian scenario, it will be very difficult to follow Mediterranean diet, so a concept of Indo-Mediterranean was diet was introduced in a study by Singh et al. Total 499 patients were allocated to a Indo -Mediterranean diet rich in whole grains, fruits, vegetables, walnuts, and almonds. 501 controls consumed a local diet similar to the step I National Cholesterol Education Program (NCEP) prudent diet. It was seen that there was significant reduction in serum cholesterol concentration and other risk factors in both groups, but especially in the intervention diet (Indo -Mediterranean) group. Indo-Mediterranean diet was shown to reduce sudden cardiac death, Myocardial infarction, weight and BMI in Obese adults on follow up. In a study by Bharti et al, it was seen that Olive oil and Mustard oil are comparable and infact Mustard oil is suitable for Indian cooking settings, hence mustard oil can be used as instead of olive oil in Indo -Mediterranean diet. In summary, MD diet has been shown to be useful in NAFLD patients, also there is very limited data in pediatric literature about the advantages of MD in NAFLD children. The investigators aim compare the effect of Indo-Mediterranean diet and calorie restricted on hepatic steatosis and fibrosis in Overweight Indian children and adolescent with Biopsy proven NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-18 years
* BMI > 85th centile
* Ultrasonography abdomen s/o Fatty Liver
* Biopsy proven NAFLD

Exclusion Criteria:

* Other Liver diseases such as Viral hepatitis (Hep B and C), Autoimmune hepatitis, Wilson disease
* Liver Biopsy not done
* Refused Consent

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
The Primary outcome measure will be a composite end point defined by decrease in Controlled Attenuation Parameter (CAP) and Alanine Aminotransferase (ALT) values by 10% from baseline and decrease in Pediatric NAFLD Fibrosis Index score <3 | 180 days
  Decrease in CAP and ALT values by 10% from baseline and decrease in Pediatric NAFLD Fibrosis Index score <3

SECONDARY OUTCOMES:
Weight (Time frame : Change in Weight of atleast 7% from baseline at 180 days) | 180 days
  Weight will be recorded at the baseline and at the completion of diet intervention
Lipid Profile (Time frame : Change in Cholesterol, triglycerides of atleast 10% from baseline at 180 days) | 180 days
  Lipid profile will be measured in a fasting state

CONTACTS AND LOCATIONS:
Overall Officials: Aniket Deshmukh, DM, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of liver and biliary sciences, Delhi, India

REFERENCES:
- [Derived] Deshmukh A, Sood V, Lal BB, Khanna R, Alam S, Sarin SK. Effect of Indo-Mediterranean diet versus calorie-restricted diet in children with non-alcoholic fatty liver disease: A pilot randomized control trial. Pediatr Obes. 2024 Nov;19(11):e13163. doi: 10.1111/ijpo.13163. Epub 2024 Sep 2. PMID 39223952